CLINICAL TRIAL: NCT05461807
Title: Effectiveness and Safety of Rivaroxaban Compared With Apixaban in Cancer-Associated Venous Thromboembolism: A Head-to-Head (H2H) Analysis of the United States Cohort of the Observational Study in Cancer Associated Thrombosis for Rivaroxaban (H2H-OSCAR-US)
Brief Title: An Observational Study Called H2H-OSCAR-US to Learn More About How Well Rivaroxaban Works and How Safe it is Compared to Apixaban Under Real World Conditions in People in the US With Cancer Who Have Problems Due to Formation of Blood Clots in the Veins (Venous Thromboembolism)
Acronym: H2H-OSCAR-US
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 22290
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Treatment of Venous Thromboembolism in Cancer Patients; Venous Thromboembolism; Cancer
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with venous thromboembolism (VTE): Adults diagnosed with active (primary or metastatic) cancer excluding oesophageal, gastric, unresected colorectal, bladder, central nervous system cancers (except brain) and leukaemia (a cohort of CAT (Cancer-associated thrombosis) patients at a low risk for bleeding, which is defined as per the ISTH (International Society on Thrombosis and Haemostasis) guidelines), admitted to the hospital, emergency department or observation unit for acute DVT (Deep vein thrombosis) and/or PE (Pulmonary embolism) on or after January 1, 2013 (to correspond with the US availability of rivaroxaban for VTE treatment), being treated with a therapeutic VTE dose of rivaroxaban or apixaban on day 7 post-acute VTE diagnosis (index date).
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Apixaban

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Retrospective cohort analysis using United States Optum De-Identified Electronic Health Records data
Drug: Apixaban — Retrospective cohort analysis using United States Optum De-Identified Electronic Health Records data

SUMMARY:
This is an observational study in which patient data from the past on venous thromboembolism (VTE) in people with cancer is studied. In observational studies, only observations are made without specified advice or interventions.

People with VTE have problems due to the formation of blood clots in the veins. Blood clots can reduce the flow of blood to vital organs such as the lungs, which can lead to their damage. VTE can also be "recurrent". This means that the blood clots have returned after treatment. People who have cancer are more likely to develop VTE, recurrent clots, and bleeding on blood thinning treatments.

To prevent the formation of new or recurrent clots in people with cancer, a newer type of blood thinner is available, called direct-acting oral anticoagulant (DOAC). Rivaroxaban and apixaban are the most used DOACs in the US. They work by blocking a certain step in the blood clotting process, the activation of a protein called Factor X.

Previous studies show that DOACs may reduce clot risk compared to other available treatments but may potentially lead to more frequent bleeding. Studies looking at these points in direct comparison of rivaroxaban and apixaban a currently missing.

Therefore, this study will collect real-world data from the US to learn how well rivaroxaban works and how safe it is compared to apixaban in people with cancer and VTE who are at low risk for bleeding.

To do this, researchers will look at the proportion of patients that will develop:

* recurrent blood clots in the veins after treatment
* bleeding in a critical organ
* bleeding that requires a hospital stay within 3 and 6 months after participants had a VTE that was treated with rivaroxaban or apixaban.

De-identified data collected will cover 12 months before and at maximum 6 months after this VTE. They will come from US electronic health records and will cover the years 2012 to 2020.

No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age at the time of anticoagulation initiation.
* Have active cancer defined as cancer being actively treated, diagnosed within 6-months prior of the index CAT or associated with metastatic disease (regardless of time from initial cancer diagnosis)
* Admitted to the hospital, emergency department or observation unit for acute Deep vein thrombosis (DVT) and/or Pulmonary embolism (PE)
* Started on a therapeutic VTE dose of rivaroxaban or apixaban within 7 days of the qualifying VTE event and treated with a therapeutic VTE dose of rivaroxaban or apixaban as their first anticoagulant on day 7 post-acute CAT event diagnosis (index date) to increase the probability of accurately classifying patients' intended outpatient anticoagulant for CAT treatment, and that, patients are compared at the same point from diagnosis.
* Have been active in the data set for at least 12-months prior to the index event (based on the "First Month Active" field) and had at least one provider visit in the 12-months prior to the acute VTE event (baseline period).

Exclusion Criteria:

* Oesophageal, gastric, unresected colorectal, bladder, central nervous system cancers (except brain) and leukaemia
* Evidence of atrial fibrillation, recent hip/knee replacement (within 35 days of index VTE), ongoing VTE treatment, valvular heart disease defined as any rheumatic heart disease, mitral stenosis, or mitral valve repair/replacement.
* Pregnancy.
* Initiation of non-therapeutic VTE doses of rivaroxaban or apixaban.
* Evidence of anticoagulation use written prescription or patient self-report during the 12-months prior to the qualifying CAT event per.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with active (primary or metastatic) cancer excluding oesophageal, gastric, unresected colorectal, bladder, central nervous system cancers (except brain) and leukaemia (a cohort of CAT patients at a low risk for bleeding, which is defined as per ISTH guidelines), experiencing a hospital, emergency department, or observation unit admission with a primary diagnosis code for VTE, who received therapeutic VTE doses of rivaroxaban or apixaban as their first outpatient anticoagulant (index event) within 7-days of the acute VTE event and were active in the data set for at least 12-months prior to the CAT event and with at least one provider visit in the 12-months prior to the acute CAT event (establishing a 12-month look back/baseline period).
Sampling Method: Non-Probability Sample
Enrollment: 2437 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Composite of recurrent VTE (fatal and non-fatal) or any bleed resulting in hospitalization (per the Cunningham algorithm) at 3 months | Retrospective data analysis from January,2013 to December,2020
Composite of recurrent VTE (fatal and non-fatal) or any critical organ bleed (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, or pericardial, or intramuscular with compartment syndrome) at 3 months | Retrospective data analysis from January,2013 to December,2020
Recurrent VTE (fatal and non-fatal) at 3 months | Retrospective data analysis from January,2013 to December,2020
Any bleed resulting in hospitalization (per the Cunningham algorithm) at 3 months | Retrospective data analysis from January,2013 to December,2020
Critical organ bleeding (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, or pericardial, or intramuscular with compartment syndrome) at 3 months | Retrospective data analysis from January,2013 to December,2020

SECONDARY OUTCOMES:
Composite of recurrent VTE (fatal and non-fatal) or any bleed resulting in hospitalization (per the Cunningham algorithm) at 6 months | Retrospective data analysis from January,2013 to December,2020
Composite of recurrent VTE (fatal and non-fatal) or any critical organ bleed (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, or pericardial, or intramuscular with compartment syndrome) at 6 months | Retrospective data analysis from January,2013 to December,2020
Recurrent VTE (fatal and non-fatal) at 6 months | Retrospective data analysis from January,2013 to December,2020
Any bleed resulting in hospitalization (per the Cunningham algorithm) at 6 months | Retrospective data analysis from January,2013 to December,2020
Critical organ bleeding (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, or pericardial, or intramuscular with compartment syndrome) at 6 months | Retrospective data analysis from January,2013 to December,2020

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Wuppertal, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Caroti KS, Becattini C, Carrier M, Cohen AT, Ekbom A, Khorana AA, Lee AYY, Brescia C, Abdelgawwad K, Psaroudakis G, Rivera M, Schaefer B, Brobert G, Coleman CI. Rivaroxaban versus Apixaban for Treatment of Cancer-Associated Venous Thromboembolism in Patients at Lower Risk of Bleeding. TH Open. 2023 Jul 10;7(3):e206-e216. doi: 10.1055/s-0043-1770783. eCollection 2023 Jul. PMID 37435565